CLINICAL TRIAL: NCT03361280
Title: Beta-blocker Dialyzability in Maintenance Hemodialysis Patients
Brief Title: Removal of Beta Blocker Drugs by Hemodialysis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 104909
Record Dates: First submitted 2017-11-21; First posted 2017-12-04 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Chronic Kidney Diseases
Keywords: hemodialysis; dialytic clearance; pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Adrenergic beta-Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Atenolol (Experimental): Atenolol (50 mg) administered 3 hours prior to a hemodialysis session. Blood samples are collected a multiple times during dialysis and spent dialysate is collected at the end of the dialysis session.
  Interventions: Drug: Beta blocker
- Bisoprolol (Experimental): Bisoprolol (5 mg) administered 3 hours prior to a hemodialysis session. Blood samples are collected a multiple times during dialysis and spent dialysate is collected at the end of the dialysis session.
  Interventions: Drug: Beta blocker
- Metoprolol (Experimental): Metoprolol (50 mg) administered 3 hours prior to a hemodialysis session. Blood samples are collected a multiple times during dialysis and spent dialysate is collected at the end of the dialysis session.
  Interventions: Drug: Beta blocker
- Carvedilol (Experimental): Carvedilol (6.25 mg) administered 3 hours prior to a hemodialysis session. Blood samples are collected a multiple times during dialysis and spent dialysate is collected at the end of the dialysis session.
  Interventions: Drug: Beta blocker

INTERVENTIONS:
Drug: Beta blocker — Beta blockers are administered as described in arms.

SUMMARY:
Eight maintenance hemodialysis patients are given one of four beta blocker drugs (atenolol, bisoprolol, carvedilol, metoprolol) three hours prior to a hemodialysis session. Blood samples and spent dialysate are collected during dialysis. On separate dialysis sessions, patients received the other study drugs until they have taken each of the four study drugs. Dialytic clearance is calculated.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age, receiving hemodialysis three times per week for at least 90 days.

Exclusion Criteria:

* gastrointestinal or liver disease, body mass index greater than 40 kg/m2, contraindications for receiving a beta blocker (treatment with contraindicated medications, prior adverse reaction, severe reactive airway disease, hemodynamic instability during dialysis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-02-27 (Actual); Primary Completion 2016-03-10 (Actual); Study Completion 2016-03-10 (Actual)

PRIMARY OUTCOMES:
Dialytic Clearance | Through study completion, average of one year.
  Dialytic clearance calculated by the recovery clearance method

SECONDARY OUTCOMES:
Dialytic Clearance | Through study completion, average of one year.
  Dialytic clearance calculated by the arteriovenous difference method

IPD SHARING:
Plan to Share IPD: No
Plasma concentrations of beta blockers will be shared with other researchers if requested.